CLINICAL TRIAL: NCT03954769
Title: A Pilot Study of the Psychometric Properties of the "Stanford Proxy Test for Delirium" (S-PTD): a New Screening Tool for the Detection of Delirium
Brief Title: A Pilot Study of "Stanford Proxy Test for Delirium" (S-PTD)
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jose R Maldonado, MD, Associate Professor, Stanford University
Other Study IDs: 28327
Record Dates: First submitted 2014-04-14; First posted 2019-05-17 (Actual); Last update posted 2019-05-17 (Actual); Status verified 2019-04

CONDITIONS: Hyperactive Delirium; Hypoactive Delirium; Mixed Type Delirium
Keywords: Delirium,; Confusion Assessment Method; Proxy Test of Delirium; DSM-V; Hyperactive Delirium; Hypoactive Delirium; Mixed-type delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Inpatients: Patients admitted to Stanford Hospital and Clinics medical and surgical units

SUMMARY:
Although there are several tools available for the screening of delirium among the medically ill, they all have some limitations. First, none of the available tools have been validated against newly developed and published DSM-5 (Diagnostic and Statistical Manual) or ICD-10 (International Statistical Classification of Diseases and Related Health Problems) criteria. Additionally, all the screening/diagnostic tools presently available have the same limitation, they all require significant patient involvement and participation (e.g., questions and activities) in order to complete the assessment. By definition, delirium is a neuropsychiatric disorder characterized by disturbance in attention and awareness, and additional disturbance in cognition (e.g., memory deficit, disorientation), language, visuospatial ability, or perception. The intrinsic characteristics of delirium seem to interfere with the patient's ability to participate and complete many of the tasks associated with delirium evaluation itself. Finally, most available tools seem to narrowly focus on some neurocognitive areas of delirium, but not being comprehensive enough.

In contrast, the S-PTD is designed so it can be completed by the nursing staff caring for the patients, the medical personnel most intimately involved with the care and aware of the behaviors exhibited by the patient during the course of their hospital stay. The idea is that nurses will complete the screening tool (hence the term "by proxy"), based on the behaviors and interactions observed during the course of a conventional "nursing shift", to determine whether the patient meets current neuropsychiatric criteria for the diagnosis of delirium.

DETAILED DESCRIPTION:
Patients admitted to Stanford Hospital and Clinics medical and surgical units meeting the study's inclusion and exclusion criteria will be considered for enrollment during the recruitment phase.

The research personnel, under the supervision of the study PI (an expert in delirium), will perform daily study procedures as follows:

A member of the research team will obtain a list of all newly admitted patients from the prior 24 hours each Monday through Friday morning from the unit's nurse manager. A member of the research team will also look at daily operating room schedules for patients to be admitted to participating units post-operatively, having received permission to do so from the directors of participating medical/surgical services. Given that the purpose of this tool is to screen for a condition that may occur in medically ill patients, every newly admitted patient or their surrogate (for those lacking decisional making capacity), meeting inclusion criteria will be approached for participation in the study and asked to provide consent. Patients lacking capacity for consent will not be automatically excluded, given that the inclusion of delirious patients is critical for adequate evaluation of the S-PTD, and most delirious patients, by definition, lack capacity to provide informed consent. We will ask for the consent from surrogate decision makers in these cases.

In addition, it is anticipated that some patients who meet eligibility will be unable to sign a consent form due to physical limitations related to their hospitalization (e.g. patients recovering from recent surgery). If a patient is unable to sign the consent form due to physical limitations, oral consent will be obtained. Oral consent will also be used in the event that a patient lacks capacity and has no surrogate decision-maker at bedside, but a surrogate decision-maker is available by phone. For Spanish-speaking patients, consent will be obtained by the same procedures utilizing Spanish-language written/oral consent, with the help of SHC interpreter services.

For each patient that consents to participate in the study, the nurse assigned to that patient during the shift will be approached. These nurses will additionally be asked to provide consent, as they are also subjects of the study.

All patients will be followed for the duration of their hospital stay (expected to average 5 days), to a maximum of two weeks, except in the case of delirious patients, who will be followed until the resolution of the episode of delirium.

Every day, enrolled patients will undergo two, separate evaluations. Towards the end of their shift (within the last 2-hrs of each shift) the patient's nurse will complete the S-PTD, utilizing all available data from the entire nursing shift (8-12 hours, depending the unit's shift mode), which allows nurses to take into account all of nurse's interactions and observations across the entire shift (including direct interactions between the patient and the nurse, family and all clinical staff). In addition, patients will undergo a clinical neuropsychiatric examination performed by a neuropsychiatrist (the gold standard), estimated to take about 5 minutes. The examiners will be blind to the results of each other's exam. Finally, a member of the research team, blind to the results of the previous tests, will conduct a separate interview of the patient's nurse towards the end of the shift in order collect the nurse's forms and evaluate the nurse's opinions regarding the ease to complete the S-PTD.

Later the results of the S-PTD will be compared against the results of the neuropsychiatric examination. The sensitivity, specificity, positive predictive value, and negative predictive value of the S-PTD will be calculated as compared to the results of clinical neuropsychiatric evaluation based on DSM-5 criteria.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for enrolled patients:

  * all inpatients admitted to Stanford Hospital's selected general medical and surgical units
  * patients must be able to communicate and read English and/or Spanish
  * ages 18 and older
* Inclusion criteria for enrolled nurses:

  * All nurses assigned to each enrolled patient for the shift during which that patient is enrolled, will be invited to participate in the study to assess the tool's acceptability and ease of use.

Exclusion Criteria:

* For enrolled patients:

  * unable to speak English or Spanish.
  * unwillingness to participate in the study
  * for patients who are unable to consent (i.e., lack capacity), either the lack of availability of a suitable surrogate or the surrogate's unwillingness to provide consent
* For enrolled nurses: unwillingness to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to selected Stanford Hospital and Clinics general medical/surgical units, for any diagnosis. Both female and male patients, English or Spanish-speaking subjects, age 18 and above, of any ethnic background will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Incidence of delirium | The study will be carried out over a 2-year period; patients will be followed throughout the hospital stay, for a maximum of 2-weeks from the time of admission, or until discharge.
  Every day, enrolled patients will undergo two evaluations: (1) At the end of the nursing shift, nurses will complete the S-PTD based on the entirety of the interactions with the patient throughout the course of their shift, estimated to take about 2-3 minutes; (2) then, within 1-hour of the nurse's S-PTD assessment a member of the Psychosomatic Medicine Service will conduct a blinded clinical neuropsychiatric examination (the gold standard for delirium diagnosis). At the end of their nursing shift (either 8 or 12 hours).

CONTACTS AND LOCATIONS:
Overall Officials: Jose R Maldonado, M.D., Principal Investigator — Stanford University
Locations (1):
- Stanford Hospital and Clinics, Stanford, California, United States

REFERENCES:
- [Background] Maldonado JR. Delirium in the acute care setting: characteristics, diagnosis and treatment. Crit Care Clin. 2008 Oct;24(4):657-722, vii. doi: 10.1016/j.ccc.2008.05.008. PMID 18929939
- [Background] Siddiqi N, House AO, Holmes JD. Occurrence and outcome of delirium in medical in-patients: a systematic literature review. Age Ageing. 2006 Jul;35(4):350-64. doi: 10.1093/ageing/afl005. Epub 2006 Apr 28. PMID 16648149
- [Background] Ryan DJ, O'Regan NA, Caoimh RO, Clare J, O'Connor M, Leonard M, McFarland J, Tighe S, O'Sullivan K, Trzepacz PT, Meagher D, Timmons S. Delirium in an adult acute hospital population: predictors, prevalence and detection. BMJ Open. 2013 Jan 7;3(1):e001772. doi: 10.1136/bmjopen-2012-001772. PMID 23299110
- [Background] Norbaek J, Glipstrup E. Delirium is seen in one-third of patients in an acute hospital setting. Identification, pharmacologic and non-pharmacologic treatment is inadequate. Dan Med J. 2016 Nov;63(11):A5293. PMID 27808035